CLINICAL TRIAL: NCT06672952
Title: Dose-Response Impact of Glucosyl-Hesperidin (CitraPeak) on Exercise Performance, Blood Flow, Stress, Cognition, and Other Perceptual Indicators
Acronym: HES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lindenwood University (Other)
Collaborators: Increnovo, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB-24-82
Record Dates: First submitted 2024-11-01; First posted 2024-11-04 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Exercise Performance; Exercise Recovery; Cognitive Function; Nitric Oxide; Blood Flow; Endurance Exercise
Keywords: exercise performance; aerobic capacity; anaerobic power; mood; nitric oxide; cognitive function; glucosyl-hesperidin; training readiness; fuel utilization; endothelial function
MeSH Terms: interventions — glucosyl hesperidin; Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This study employs a double-blind design to ensure that participants, investigators, and outcome assessors remain unaware of the group assignments. All supplements (placebo and both doses of CITRAPEAK®) are provided in identical capsules, containing either 400 mg of cellulose (placebo), 200 mg of CITRAPEAK® with 200 mg of cellulose, or 400 mg of CITRAPEAK®. Each participant is assigned a unique randomization code, which is used to label the capsules, maintaining blinding throughout the study. Only the study designated unblinded personnel have access to the randomization key, ensuring that the blinding remains intact for all other study staff.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Participants in this arm will receive a placebo supplement consisting of 400 mg of cellulose per day. The placebo is designed to match the appearance and dosage form of the active interventions, allowing for blinding in the study.
  Interventions: Dietary Supplement: Placebo
- 200 mg CITRAPEAK® (glucosyl-hesperidin) supplementation (Experimental): Participants in this arm will receive a total of 200 mg of glucosyl-hesperidin (CITRAPEAK®) supplementation per day, along with an additional 200 mg of cellulose. This will provide a daily dosage of 400 mg, maintaining blinding to ensure the placebo effect is accounted for.
  Interventions: Dietary Supplement: 200 mg CITRAPEAK® (glucosyl-hesperidin) supplementation
- 400 mg CITRAPEAK® (glucosyl-hesperidin) supplementation (Experimental): Participants in this arm will receive a total of 400 mg of glucosyl-hesperidin (CITRAPEAK®) supplementation per day. This higher dose is intended to evaluate its effects on exercise performance, recovery, and cognitive function compared to the placebo and lower dose.
  Interventions: Dietary Supplement: 400 mg CITRAPEAK® (glucosyl-hesperidin) supplementation

INTERVENTIONS:
Dietary Supplement: 400 mg CITRAPEAK® (glucosyl-hesperidin) supplementation — The active intervention consists of 400 mg of glucosyl-hesperidin (CITRAPEAK®) in capsule form.
  Arms: 400 mg CITRAPEAK® (glucosyl-hesperidin) supplementation
Dietary Supplement: Placebo — The placebo intervention consists of 400 mg/day of cellulose in capsule form, matching the appearance and dosage of active interventions.
  Arms: Placebo
Dietary Supplement: 200 mg CITRAPEAK® (glucosyl-hesperidin) supplementation — The active intervention includes 200 mg of glucosyl-hesperidin (CITRAPEAK®) and an additional 200 mg of cellulose in capsule form.
  Arms: 200 mg CITRAPEAK® (glucosyl-hesperidin) supplementation

SUMMARY:
The purpose of this study is to evaluate the dose-dependent effects of glucosyl-hesperidin (CITRAPEAK) supplementation on exercise performance, recovery indicators, blood flow, cognitive function, mood, sleep, and fuel utilization in recreationally active adults.

DETAILED DESCRIPTION:
This randomized, double-blind, placebo-controlled study investigates the effects of glucosyl-hesperidin (CITRAPEAK) on exercise performance, recovery, cognitive function, mood, and cardiovascular health in approximately 60 healthy, recreationally active adults aged 18-50. Participants will be assigned to one of three groups (placebo, 200mg CITRAPEAK, or 400mg CITRAPEAK) based on sex and baseline fat-free mass. Each participant will consume their assigned supplement daily for 8 weeks, with adherence tracked via supplementation logs. The study includes multiple visits, where participants will undergo a range of assessments, including exercise performance tests, blood flow analysis, and cognitive evaluations.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who are between 18 - 50 years of age
2. Body mass index values will range from >25.0 < 30.0 kg/m2
3. The average body mass index for entire study cohort will be less than 27.0 kg/m2. As such an ongoing calculation of the recruited cohort's mean body mass index will be maintained and people will only be randomized into the study if the average cohort body mass index value does not exceed 27.0 kg/m2
4. Free-living and independent
5. In good health absent of being overweight or mildly obese with no other signs or symptoms of cardiovascular, respiratory, metabolic, immune, psychiatric, or musculoskeletal disease or disorders
6. Willingness to maintain consistent sleep duration the evening before study visits
7. Willing and able to agree to the requirements and restrictions of this study, be willing to give voluntary consent, and carry out all study-related procedures
8. Regular completion of at least 180 minutes of moderate to vigorous exercise per week for the past 6 months

Exclusion Criteria:

1. Not currently completing at least 180 minutes of moderate to vigorous exercise per week for the past 6 months
2. Positive medical history and/or is currently being treated for some form of heart disease, cardiovascular disease
3. Currently being treated for kidney disease, renal failure, or has dialysis performed on regular intervals
4. Has liver disease or some form of clinically diagnosed hepatic impairment
5. Diagnosed with having Type I or Type II diabetes (determined as fasting blood glucose > 126 mg/dL)
6. Diagnosed with or is being treated for some form of thyroid disease
7. Diagnosed with major affective disorder or other psychiatric disorder that required hospitalization in the prior year
8. Diagnosed with some form of immune disorder (i.e., HIV/AIDS)
9. History of cancer (except localized skin cancer without metastases or in situ cervical cancer within 5 years prior to screening visit).
10. Participant has an abnormality or obstruction of the gastrointestinal tract precluding swallowing (e.g., dysphagia) and digestion (e.g., known intestinal malabsorption, celiac disease, inflammatory bowel disease, chronic pancreatitis, steatorrhea)
11. Positive medical history for any neurological condition or neurological disease
12. Currently prescribed a statin drugs (i.e., Lipitor, Livalo, Crestor, Zocor, etc.) or any hypertension medications (i.e., Beta-blockers, ACE Inhibitors, Alpha blockers, Vasodilators, etc.)
13. Current smoker (average of > 1 pack per day within the past 3 months) has quit within the past six months. This includes all forms of nicotine
14. Intake of any drugs (prescribed or over the counter) or dietary supplements that are known or are purported to weight loss such as thermogenics, hydroxycitric acid, ephedra, capsaicin, etc.
15. Participants who are lactating, pregnant or planning to become pregnant
16. Have a known sensitivity or allergy to any of the study products
17. History of alcohol or substance abuse in the 12 months prior to screening
18. Receipt or use of an investigational product in another research study within 30 days of beginning the study protocol
19. Any orthopedic limitation that would prevent participation in a general fitness program
20. Any condition or abnormality that, in the opinion of the investigator, would compromise the safety of the participant or the quality of the study data

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Peak VO2 at Week 8 Following Glucosyl-Hesperidin (CITRAPEAK) Supplementation | Baseline and Week 8
  Peak VO2 will be measured as an indicator of maximal aerobic capacity. Higher values reflect improved cardiovascular performance.
Change from Baseline in Wingate Anaerobic Test Peak Anaerobic Power at Week 8 Following Glucosyl-Hesperidin (CITRAPEAK) Supplementation | Baseline and Week 8
  Peak anaerobic power will be measured to assess maximal power output during high-intensity exercise. Higher values indicate improved anaerobic performance.
Change from Baseline in Wingate Anaerobic Test Mean Anaerobic Power at Week 8 Following Glucosyl-Hesperidin (CITRAPEAK) Supplementation | Baseline and Week 8
  Wingate Anaerobic Test Mean anaerobic power will be recorded during repeated high-intensity exercise, with higher values indicating enhanced anaerobic endurance.
Change from Baseline in Fatigue Rate at Week 8 Following Glucosyl-Hesperidin (CITRAPEAK) Supplementation | Baseline and Week 8
  Wingate Anaerobic Test Fatigue rate will be measured as the decline in power over time during anaerobic exercise, with a lower rate indicating improved endurance.
Change from Baseline in Perceived Indicators of Recovery, Training Readiness, Soreness, and Overall Feel Using Visual Analog Scales (VAS) at Week 8 Following Glucosyl-Hesperidin (CITRAPEAK) Supplementation | Baseline and Week 8
  Perceived recovery, training readiness, soreness, recovery, and general "feel" will be self-rated using visual analog scales (VAS), with higher values indicating greater perceived improvements in each category.
Change from Baseline in Brachial Artery Blood Flow Measured 0, 30, and 60 Minutes After Acute and Prolonged Ingestion of Glucosyl-Hesperidin (CITRAPEAK) | Baseline and Week 8, measured at 0, 30, and 60 minutes post-ingestion.
  Brachial artery blood flow will be measured to assess vascular response to CITRAPEAK at baseline and after 8 weeks of supplementation, with measurements taken at 0, 30, and 60 minutes post-ingestion.

SECONDARY OUTCOMES:
Change from Baseline in Carbohydrate and Fat Oxidation Rates at 30%, 40%, 50%, 60%, 70%, and 80% Peak VO2 During Exercise at Week 8 Following Glucosyl-Hesperidin (CITRAPEAK) Supplementation | Baseline and Week 8
  Carbohydrate and fat oxidation rates will be measured at incremental intensities to assess fuel utilization during exercise, with higher fat oxidation indicating improved metabolic flexibility.
Change from Baseline in Stroop Color Matching Test Performance 0, 30, and 60 Minutes After Ingesting Dose 1 (Week 0) and Dose 56 (Week 8) Following Glucosyl-Hesperidin (CITRAPEAK) Supplementation | 0, 30, and 60 minutes post-ingestion at baseline and Week 8
  The Stroop color matching test will be conducted to assess cognitive processing speed and accuracy. Testing will occur at 0, 30, and 60 minutes after ingestion of the initial dose (Week 0) and the final dose (Week 8). Improved scores indicate enhanced cognitive performance.
Change from Baseline in Trail Making Test Performance 0, 30, and 60 Minutes After Ingesting Dose 1 (Week 0) and Dose 56 (Week 8) Following Glucosyl-Hesperidin (CITRAPEAK) Supplementation | 0, 30, and 60 minutes post-ingestion at baseline and Week 8
  The Trail Making Test will be conducted to evaluate cognitive flexibility and executive function. Testing will occur at 0, 30, and 60 minutes after ingestion of the initial dose (Week 0) and the final dose (Week 8). Faster completion times indicate improved cognitive function.
Change from Baseline in Profile of Mood States (POMS) Score at Week 8 Following Glucosyl-Hesperidin (CITRAPEAK) Supplementation | Baseline and Week 8
  The Profile of Mood States (POMS) questionnaire will assess mood states across several domains, with lower scores indicating improved mood and well-being.
Change from Baseline in Pittsburgh Sleep Quality Index (PSQI) Score at Week 8 Following Glucosyl-Hesperidin (CITRAPEAK) Supplementation | Baseline and Week 8
  The Pittsburgh Sleep Quality Index (PSQI) will assess subjective sleep quality, with lower scores reflecting better sleep.
Change from Baseline in Plasma Nitric Oxide Levels at Week 8 Following Glucosyl-Hesperidin (CITRAPEAK) Supplementation | Baseline and Week 8
  Plasma nitric oxide levels will be measured to evaluate changes in endothelial function, with higher levels suggesting improved vasodilation.

CONTACTS AND LOCATIONS:
Overall Officials: Chad M Kerksick, PhD, Principal Investigator — Lindenwood University
Locations (1):
- Lindenwood University, Saint Charles, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan to share IPD